CLINICAL TRIAL: NCT00915655
Title: A Phase II, Open-Label Trial, to Evaluate Pharmacokinetics, Safety, Tolerability and Antiviral Activity of Drv/Rtv Once Daily in Treatment-Naive HIV-1 Infected Adolescents Aged Between 12 and < 18 Years
Brief Title: A Study to Evaluate Antiviral Activity of Darunavir + Ritonavir in HIV-1 Infected Adolescents
Acronym: DIONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016312; TMC114-TiDP29-C230 (Other: Tibotec Pharmaceuticals, Ireland); 2008-004631-37 (EudraCT Number)
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2011-12-28 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: HIV-1 Infection
Keywords: HIV Infections; TMC114-TiDP29-C230; TMC114-C230; TMC114; HIV-1; Darunavir; Ritonavir; NRTI; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; Zidovudine; Lamivudine; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DRV/rtv (darunavir/ritonavir) (Experimental): Patients will receive darunavir tablets 2 x 400 mg in combination with ritonavir capsule 100 mg once daily for 48 weeks along with 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) ie, either zidovudine/lamivudine or abacavir/lamivudine
  Interventions: Drug: darunavir; Drug: ritonavir; Drug: zidovudine; Drug: lamivudine; Drug: abacavir

INTERVENTIONS:
Drug: darunavir — Type=exact number, unit=mg, number=400, formulation=tablet, route=oral. 2 tablets of darunavir administered once daily for 48 weeks
  Other Names: DRV
Drug: ritonavir — Type=exact number, unit=mg, number=100, formulation=capsule, route=oral. 1 capsule of ritonavir administered once daily for 48 weeks
  Other Names: rtv
Drug: zidovudine — NRTI (zidovudine) administered as per approved, marketed, or considered local standard of care for patients aged between 12 and < 18 years in a particular country
Drug: lamivudine — NRTI (lamivudine) administered as per approved, marketed, or considered local standard of care for patients aged between 12 and < 18 years in a particular country
Drug: abacavir — NRTI (abacavir) administered as per approved, marketed, or considered local standard of care for patients aged between 12 and < 18 years in a particular country

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics (what body does to medication), safety, tolerability, and efficacy (effectiveness) of darunavir with low-dose ritonavir (DRV/rtv) administered once daily, in combination with an investigator-selected background regimen consisting of other antiretrovirals (ARVs) ie, 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs), in treatment-naive (never treated before) HIV-1 infected adolescents aged from 12 to <18 years and weighing at least 40 kg.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-arm, Phase II study to evaluate the pharmacokinetics, safety, tolerability, and efficacy of darunavir/ritonavir (DRV/rtv) administered once daily, in combination an investigator-selected background regimen (2 NRTIs), in treatment-naive HIV-1 infected adolescents over 48 weeks. A total of 12 patients will be enrolled in this study. Patients will be considered treatment-naive if they have never received treatment with an ARV medication, including both investigational as well as commercially available ARVs indicated for the treatment of HIV-infection and ARVs for the treatment of hepatitis B infection with anti-HIV activity. The investigator-selected background regimen will consist of 2 NRTIs, either zidovudine/lamivudine or abacavir/lamivudine, whichever is approved and marketed or considered local standard of care for adolescents aged from 12 to <18 years in a particular country. The study will consist of a 4-week screening period, a 48-week treatment period, and a 4-week follow-up period. Safety, efficacy, resistance (reduction in effectiveness of a medication), pharmacokinetic analyses, and pharmacodynamic (what medication does to body) analyses will be performed at Week 24 (primary analysis) and Week 48 (final analysis). Patients who will complete the 48 weeks of treatment with DRV/rtv and who will continue to benefit from this treatment, will have the opportunity to continue this treatment until they no longer benefit from the medication, until DRV is commercially available or can be accessed from another source (eg, access program, government program) or until the development program is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented HIV-1 infection
* Body weight from at least 40 kg at screening
* Screening plasma HIV-1 RNA >= 1000 copies/mL
* Parents or legal representative and trial patients (where appropriate, depending on age and local regulation) willing and able to give consent and assent
* General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial
* Able to swallow darunavir tablets (400 mg) and ritonavir capsules (100 mg)

Exclusion Criteria:

* Patients with presence of any currently active conditions included in the listing of World Health Organisation (WHO) Clinical Stage 4
* Any condition (including, but not limited to, alcohol and drug use), which, in the opinion of the investigator, could compromise the patient's safety or adherence to the trial protocol
* Previous or current use of antiretrovirals (ARVs)
* Primary or acute HIV infection
* Use of any investigational agents within 30 days prior to screening
* Use of disallowed concomitant therapy
* Pregnant or breast-feeding
* Female patient of childbearing potential without use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period
* Patients with clinical or laboratory evidence of significantly decreased hepatic function or decompensation (ie, liver insufficiency), irrespective of liver enzyme levels
* Any active clinically significant disease (eg, cardiac dysfunction, pancreatitis, acute viral infection) or findings during screening of medical history or physical examination that are expected to compromise the patient's safety or outcome in the trial

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (9):
- Memphis, Tennessee, United States
- Paris, France
- Dublin, Ireland
- Spain (2):
  - Esplugues de Llobregat
  - Madrid
- Kiev, Ukraine
- United Kingdom (3):
  - Birmingham
  - Bristol
  - Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Groups:
- DRV/Rtv: Darunavir tablets 2 x 400 mg tablet once daily for 48 weeks. Ritonavir capsule 100 mg capsule once daily for 48 weeks.
Period: Overall Study
Arm/Group | DRV/Rtv
Started | 12
Completed | 12 ('Completed' represents patients who have not discontinued at time of cut-off for Week 24 analysis)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Percentile for Height [Median (Full Range); unit: Height Percentile] | 27.2 [0.5 to 94.1]
Percentile for BMI [Median (Full Range); unit: BMI Percentile] | 47.5 [13.3 to 85.9]
Percentile for Weight [Median (Full Range); unit: Weight Percentile] | 51.6 [8.6 to 79.0]

OUTCOME MEASURES:

1. Primary Outcome: Virological Response[Viral Load <50 Copies/mL, TLOVR]
Description: The analysis is based on virologic response defined as percentage of patients with confirmed plasma viral load <50 HIV-1 RNA copies/mL at Week 24 calculated according to the Food and Drug Administration (FDA) Time to Loss of Virologic Response (TLOVR) algorithm.
Time Frame: Week 24
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 12
Participants
  Yes | 11
  No | 1

2. Secondary Outcome: Virological Response [Viral Load <50 Copies/mL, FDA-SNAPSHOT]
Description: The analysis is based on the last observed viral load (VL) data within the Week 24 window. Virologic response is defined as a VL<50 copies/mL (observed case). Virologic Failure includes a) patients who had >=50 copies/mL in the Week-24 window, b) patients who discontinued prior to Week 24 for lack or loss of efficacy, c) patients who had a switch in their background regimen that was not permitted by the protocol, and d) patients who discontinued for reasons other than adverse events (AEs)/death, and lack or loss of efficacy (provided their last available viral load was detectable).
Time Frame: Week 24
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Description: Only patients who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. patients with Non-Serious Adverse Events.
Arm/Group | DRV/Rtv
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv (N=12)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv (N=12)
Furuncle (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Asymptomatic bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Nail injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Uterine cervical erosion (Reproductive system and breast disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will not unreasonably withhold consent to publish the data generated in this trial. However, it is the policy of the Sponsor not to allow the investigators to publish their results or findings prior to the Sponsor's publication of the overall trial results. The investigator agrees that before he/she publishes any results of this trial, he/she shall allow at least 45 days for the Sponsor to review the prepublication manuscript prior to submission of the manuscript to the publisher.